CLINICAL TRIAL: NCT06602778
Title: Association of Physical Activity Level and Sleep Quality with Oxidative Stress and Exercise-related Biomarker Levels in Type 2 Diabetes
Brief Title: Physical Activity Level and Sleep Quality in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assist.Prof.Dr., Selcuk University
Other Study IDs: 2024/09.17
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Sleep; Biomarkers / Blood; Physical Activity Level
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Biomarkers; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- T2DM-BMI0
  Interventions: Other: Biomarkers / blood; Other: Questionnaire
- T2DM-BMI1
  Interventions: Other: Biomarkers / blood; Other: Questionnaire
- T2DM-BMI2
  Interventions: Other: Biomarkers / blood; Other: Questionnaire
- T2DM-BMI3
  Interventions: Other: Biomarkers / blood; Other: Questionnaire

INTERVENTIONS:
Other: Biomarkers / blood — Analysis of routine biochemical parameters
Other: Questionnaire — Physical activity level will be assessed using the International Physical Activity Questionnaire Short Form (IPQI) and sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The data to be obtained from blood will be obtained by selecting blood samples that will be sent to biological waste.

SUMMARY:
In this study, we investigated the effects of physical activity level and sleep quality level on total antioxidant level (TAS), total oxidant level (TOS), Malondialdehyde (MDA) and Superoxide Dismutase (SOD) which are markers of oxidative stress, irisin, fibronectin type III-protein 5 (FNDC5).

ELIGIBILITY:
Inclusion Criteria:

* Being between 30-65 years old
* Volunteering to participate in the study
* Being literate
* Being diagnosed with Type 2 Diabetes

Exclusion Criteria:

* Having a physical or mental illness that prevents communication
* malignant disease,
* infectious disease,
* chronic obstructive pulmonary disease,
* liver disease,
* patients with kidney disease and joint or muscle disease will not be included

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to the endocrinology department at the medical faculty hospital
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
biomarkers derived from blood sera | 10 Minutes
  blood glucose, total cholesterol, triglycerides, LDL and HDL analyzes
ELISA method of oxidative stress markers | 10 minutes
  All reagents of the ELISA kits of the oxidative stress markers TAS, TOS, MDA and SOD will be brought to room temperature. Standards will be prepared according to the protocol and added to a 96-well plate with the samples. Buffer solution will be added to each well and incubated for 90 min at room temperature. After each step, necessary washes will be performed and finally chromogenic agents will be added and read spectrophotometrically. Although the timing and additions may vary according to the parameter, in general the procedure is as indicated. Each sample will be run 2 times for both TAS and TOS
Analysis of exercise-related markers by ELISA method | 10 minutes
International Physical Activity Questionnaire | 5 minutes
Pittsburgh Sleep Quality Index | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No